CLINICAL TRIAL: NCT06091761
Title: Efficacy and Safety of Thread Embedding Acupuncture Combined With Auricular Acupuncture for Overweight and Obesity: Randomized Placebo-Controlled Trial
Brief Title: Thread Embedding Acupuncture Combined With Auricular Acupuncture for Overweight and Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Bui Pham Minh Man, Principal Investigator, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 700/HDDD-DHYD
Record Dates: First submitted 2023-10-12; First posted 2023-10-19 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Overweight or Obesity
Keywords: overweight; obesity; auricular acupuncture; thread embedding acupuncture; traditional medicine
MeSH Terms: conditions — Overweight; Obesity | interventions — Acupuncture, Ear

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will be unaware of their random allocation into either the intervention or placebo group. Sham Thread embedding acupuncture (Sham-TEA) will be administered in a manner similar to TEA, but without the insertion of threads, ensuring that no threads are left at the acupoints after the procedure.
  The physician responsible for administering the treatments will be aware of the group assignments but remain uninvolved in the evaluation of outcomes and subsequent data analysis. Those responsible for outcome assessment and data analysis will be kept blinded to the treatment assignments.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AA + TEA (Experimental): Auricular acupuncture (AA) every week in eight weeks (eight sessions). Combined with Thread embedding acupuncture (TEA) every two weeks in eight weeks (four sessions).
  Interventions: Other: Auricular acupuncture; Other: Thread embedding acupuncture
- AA + Sham-TEA (Sham Comparator): Auricular acupuncture (AA) every week in eight weeks (eight sessions). Combined with Sham Thread embedding acupuncture (Sham-TEA) every two weeks in eight weeks (four sessions).
  Interventions: Other: Auricular acupuncture; Other: Sham Thread embedding acupuncture

INTERVENTIONS:
Other: Auricular acupuncture — Auricular acupuncture is conducted weekly in eight weeks using patches, each with a square shape and a side length of 10 mm, along with sterilized needles measuring 0.25 x 1.3 mm. Five acupoints on one ear are selected, which included Shen-men (TF4), Stomach (CO4), Spleen (CO13), Endocrine (CO18), and Hunger point. The patch with the needle will remain in place for one week.
Other: Thread embedding acupuncture — Thread embedding acupuncture is performed every two weeks in eight weeks using a single Polydioxaone thread. Needles has a gauge size of 29G, a shaft length of 38mm, and a thread length of 50mm, folded in half, and are applied to ten acupoints, including Qihai (CV6), Shuifen (CV9), and Tianshu (ST25), Shuidao (ST28), Daheng (SP15), Siman (KI14) on both sides of the body. Needles with a gauge size of 30G, a shaft length of 25mm, and a thread length of 30mm, folded in half, are used for five acupoints, which included Zhongwan (CV12) and Zusanli (ST36), Pishu (BL20) on both sides of the body. After the thread being inserted into the body, the needle will be withdrawn immediately.
  Arms: AA + TEA
Other: Sham Thread embedding acupuncture — Sham Thread embedding acupuncture is performed every two weeks in eight weeks. Needles without threads has a gauge size of 29G, and a shaft length of 38mm, are applied to ten acupoints, including Qihai (CV6), Shuifen (CV9), and Tianshu (ST25), Shuidao (ST28), Daheng (SP15), Siman (KI14) on both sides of the body. Needles without threads with a gauge size of 30G, and a shaft length of 25mm, are used for five acupoints, which included Zhongwan (CV12) and Zusanli (ST36), Pishu (BL20) on both sides of the body. After the needle being inserted into the body, it will be withdrawn immediately.
  Arms: AA + Sham-TEA

SUMMARY:
Overweight and obesity are chronic non-communicable diseases with a rapidly increasing global prevalence. They constitute risk factors for various chronic conditions, including cardiovascular diseases, type 2 diabetes, chronic kidney disease, cancer, as well as musculoskeletal disorders and numerous other disorders, significantly impacting the quality of life.

Numerous non-pharmacological interventions have been employed in the management of these conditions. Particularly, Auricular acupuncture (AA) has been a widely used and established method for weight management, owing to its effectiveness, safety, and convenience. Recently, a novel therapy known as Thread embedding acupuncture (TEA) has also demonstrated efficacy in weight reduction. Several studies have shown a substantial increase in treatment effectiveness when combining TEA with other acupuncture therapies. However, there is currently no available data on the combination of TEA with AA.

This study is conducted to assess the efficacy and safety of combining TEA with AA compared with AA monotherapy in overweight and obesity.

DETAILED DESCRIPTION:
Eligible participants with overweight or obesity, defined according to the criteria set by The World Health Organization Regional Office for the Western Pacific Region (Body Mass Index [BMI] of 23 kg/m² or higher), will be enrolled and subsequently randomized into two groups: the intervention group (AA + TEA group) and the placebo group (AA + Sham-TEA group), with a 1:1 allocation ratio.

In both groups, the intervention duration is eight weeks, with Auricular acupuncture (AA) administered weekly, along with recommended lifestyle modifications. For the intervention group, Thread embedding acupuncture (TEA) therapy will be added every two weeks, totaling four sessions during the eight-week period. Meanwhile, Sham-TEA will be administered in the placebo group.

Data regarding body weight, BMI, waist circumference, hip circumference, appetite, and adverse effects will be recorded immediately following randomization and weekly thereafter over the eight-week duration.

ELIGIBILITY:
Inclusion Criteria:

* Simple overweight or obesity with a Body Mass Index (BMI) of 23 kg/m2 or higher, following the criteria of The World Health Organization Regional Office for the Western Pacific Region.
* Waist circumference of 90 cm or more for males, or 80 cm or more for females.
* Voluntary informed consent.

Exclusion Criteria:

* Secondary obesity resulting from endocrine diseases or medication.
* Presence of severe medical conditions (e.g., cardiovascular, hepatic, renal or others) that could potentially affect treatment outcomes as per researchers' assessments.
* Current use of weight-affecting medications, including diabetes medications, endocrine medications, and medications for neurological psychiatric disorders.
* Pregnancy, lactation, or recent childbirth within the past 6 months.
* Severe mental and neurological conditions that may impact treatment compliance.
* Alcohol or substance addiction.
* History of hypersensitivity reactions to any form of acupuncture with needles or to Polydioxanone.
* Existing injuries or lesions at the acupoints under investigation in this study.
* Concurrent participation in other clinical trials or utilization of other weight reduction therapies.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-03-21 (Actual); Study Completion 2024-03-21 (Actual)

PRIMARY OUTCOMES:
Changes in body weight | Assessments conducted at randomization and after each intervention week throughout the eight-week period (Week 0, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, and Week 8)
  The body weight of the participants will be collected by investigators in the morning after the participants' personal hygiene routine and before breakfast, with measurements in kilograms (kg).

SECONDARY OUTCOMES:
Changes in Body Mass Index (BMI) | Assessments conducted at randomization and after each intervention week throughout the eight-week period (Week 0, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, and Week 8)
  BMI will be calculated with the Quetelet index formula, with units in kg/m².
Changes in waist circumference | Assessments conducted at randomization and after each intervention week throughout the eight-week period (Week 0, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, and Week 8)
  The waist circumference of the participants will be measured by investigators in the morning after the participants' personal hygiene routine and before breakfast, with units in centimeters (cm).
  The waist circumference measurements will be conducted in accordance with the protocol established by the World Health Organization.
Changes in hip circumference | Assessments conducted at randomization and after each intervention week throughout the eight-week period (Week 0, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, and Week 8)
  The hip circumference of the participants will be measured by investigators in the morning after the participants' personal hygiene routine and before breakfast, with units in centimeters (cm).
  The hip circumference measurements will be conducted in accordance with the protocol established by the World Health Organization.
Changes in waist-hip ratio | Assessments conducted at randomization and after each intervention week throughout the eight-week period (Week 0, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, and Week 8)
  The waist-hip ratio will be calculated by dividing the waist circumference(cm) by the hip circumference(cm).
Changes in the Food Cravings Questionnaire-Trait-reduced (FCQ-T-r) score | Assessments conducted at randomization and after each intervention week throughout the eight-week period (Week 0, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, and Week 8)
  The FCQ-T-r consists of 15 items. Participants will be requested to express their agreement using a Likert-type scale that ranges from 1 = "strongly disagree" to 5 = "strongly agree", allowing for total scores within the range of 15 to 75, with higher scores indicating greater appetite.
Changes in Visual Analog Scale (VAS) score for appetite | Assessments conducted at randomization and after each intervention week throughout the eight-week period (Week 0, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, and Week 8)
  The VAS consists of a 100mm long line with two endpoints, ranging from "no appetite" to "greatest appetite ever experienced." Participants will mark the position on the scale that corresponds to their current appetite sensation.
Proportion of intervention-related adverse effects | Up to eight weeks
  Expected adverse events (AEs) for Auricular acupuncture include pain at the insertion site, local discomfort, local skin irritation (itching and redness), local inflammation and bleeding, chondritis, dizziness, nausea, and hypersensitivity reactions.
  For Thread embedding acupuncture, expected AEs encompass local discomfort, post-treatment elevation in body temperature, local hematoma or subcutaneous hemorrhage, local swelling, local induration, local pain, local redness, infection, abscess, pruritus, and anaphylaxis.
  Additionally, any unexpected AEs associated with these procedures will also be documented and monitored.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Medical Center HCMC - Branch no.3, Ho Chi Minh City, Vietnam

REFERENCES:
- [Background] Lillingston F, Fields P, Waechter R. Auricular Acupuncture Associated with Reduced Waist Circumference in Overweight Women-A Randomized Controlled Trial. Evid Based Complement Alternat Med. 2019 Dec 18;2019:6471560. doi: 10.1155/2019/6471560. eCollection 2019. PMID 31929817
- [Background] Yasemin C, Turan S, Kosan Z. The Effects of Auricular and Body Acupuncture in Turkish Obese Female Patients: A Randomized Controlled Trial Indicated Both Methods Lost Body Weight But Auricular Acupuncture Was Better Than Body Acupuncture. Acupunct Electrother Res. 2017 Jan;42(1):1-10. doi: 10.3727/036012917x14908026364990. PMID 29772131
- [Background] Sheng J, Jin X, Zhu J, Chen Y, Liu X. The Effectiveness of Acupoint Catgut Embedding Therapy for Abdominal Obesity: A Systematic Review and Meta-Analysis. Evid Based Complement Alternat Med. 2019 Jun 23;2019:9714313. doi: 10.1155/2019/9714313. eCollection 2019. PMID 31341504
- [Background] Wang ZY, Li XY, Gou XJ, Chen CL, Li ZY, Zhao C, Huo WG, Guo YH, Yang Y, Liu ZD. Network Meta-Analysis of Acupoint Catgut Embedding in Treatment of Simple Obesity. Evid Based Complement Alternat Med. 2022 May 23;2022:6408073. doi: 10.1155/2022/6408073. eCollection 2022. PMID 35656457
- [Background] Zhao HY, Kim S, Son MJ. Comparing acupoint catgut embedding and acupuncture therapies for simple obesity: A protocol for systematic review and meta-analysis. Medicine (Baltimore). 2022 Dec 23;101(51):e31531. doi: 10.1097/MD.0000000000031531. PMID 36595747
- [Background] Yan RH, Liu XM, Bai J, Hou BB, Yu J, Gu JS. Clinical efficacy of simple obesity treated by catgut implantation at acupoints. Chin J Integr Med. 2015 Aug;21(8):594-600. doi: 10.1007/s11655-012-1215-7. Epub 2012 Dec 3. PMID 23212565
- [Background] Wujie YE, Jingyu X, Zekai YU, Xingang HU, Yan Z. Systematic review and Meta-analysis of acupuncture and acupoint catgut embedding for the treatment of abdominal obesity. J Tradit Chin Med. 2022 Dec;42(6):848-857. doi: 10.19852/j.cnki.jtcm.2022.06.002. PMID 36378041
- [Background] Chen X, Huang W, Wei D, Zhao JP, Zhang W, Ding DG, Jiao Y, Pan HL, Zhang JJ, Zhong F, Gao F, Jin YT, Zheng YW, Zhang YJ, Huang Q, Zeng XT, Zhou ZY. Effect of Acupoint Catgut Embedding for Middle-Aged Obesity: A Multicentre, Randomised, Sham-Controlled Trial. Evid Based Complement Alternat Med. 2022 Feb 27;2022:4780019. doi: 10.1155/2022/4780019. eCollection 2022. PMID 35265146
- [Background] Jiali W, Lily L, Zhechao L, Jianping L, Mei H. Acupoint catgut embedding versus acupuncture for simple obesity: a systematic review and Meta-analysis of randomized controlled trials. J Tradit Chin Med. 2022 Dec;42(6):839-847. doi: 10.19852/j.cnki.jtcm.2022.06.001. PMID 36378040
- [Background] Dai L, Wang M, Zhang KP, Wang L, Zheng HM, Li CB, Zhou WJ, Zhou SG, Ji G. Modified acupuncture therapy, long-term acupoint stimulation versus sham control for weight control: a multicenter, randomized controlled trial. Front Endocrinol (Lausanne). 2022 Jul 28;13:952373. doi: 10.3389/fendo.2022.952373. eCollection 2022. PMID 35966092
- [Derived] Trinh DT, Kieu QV, Tran AH, Bui MP, Vuong NL. Adding thread-embedding acupuncture to auricular acupuncture enhances short-term weight reduction in overweight and obesity: A double-blinded, randomized, sham-controlled trial. Integr Med Res. 2024 Sep;13(3):101050. doi: 10.1016/j.imr.2024.101050. Epub 2024 Jun 1. PMID 38911552
- See also: Related Info — https://www.who.int/publications/i/item/9789241501491
- See also: Related Info — https://iris.who.int/handle/10665/206936?locale-attribute=es&show=full